CLINICAL TRIAL: NCT04499170
Title: Immediate Effect of the Muscle Energy Technique on Postural Control in the Elderly and Young Adults
Brief Title: Effect of Muscular Energy Technique on Postural Control
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: I left Unopar
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP07009
Record Dates: First submitted 2020-04-24; First posted 2020-08-05 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Balance Disorders Water
Keywords: Postural Balance; Musculoskeletal Manipulations; physiotherapy
MeSH Terms: interventions — Proto-Oncogene Proteins c-met

STUDY DESIGN:
Intervention Model Description: Quasi-experimental research project to detect an immediate effect of a technique on postural balance measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle energy technique (G1) (Experimental): Group Elderly (G1)
  Interventions: Other: Muscular Energy Technique G1
- Muscle energy technique (G2) (Active Comparator): Group of young people (G2)
  Interventions: Other: Muscular Energy Technique G2

INTERVENTIONS:
Other: Muscular Energy Technique G1 — Group of older (G1) - The muscular energy technique (TEM) based on Chaitow's proposal will be applied to the postural posterior muscles of the lower limbs such as gastrocnemius, soleus, ischiostibials, gluteus medius and paravertebral. During TEM, the contraction will be maintained from 7 to 10 seconds, against the resistance imposed by the therapist. After relaxation, range of motion will be gained until your new restriction barrier. This process will be repeated for 3 times.
  Other Names: "MET"
  Arms: Muscle energy technique (G1)
Other: Muscular Energy Technique G2 — Group of young people (G2) - The muscular energy technique (TEM) based on Chaitow's proposal will be applied to the postural posterior muscles of the lower limbs such as gastrocnemius, soleus, ischiostibials, gluteus medius and paravertebral. During TEM, the contraction will be maintained from 7 to 10 seconds, against the resistance imposed by the therapist. After relaxation, range of motion will be gained until your new restriction barrier. This process will be repeated for 3 times.
  Other Names: ''MET''
  Arms: Muscle energy technique (G2)

SUMMARY:
The research aims to evaluate the immediate effect of the muscle energy technique (TEM) on postural control responses in the elderly and young adults. The sample will be selected for convenience, being participants of both sexes, young and old. Evaluation of postural control through the force platform will be performed during the unipodal and semi-tandem balance tests. The main parameters of postural control will be calculated using the pressure center derivative. After the balance tests, the participants will be submitted to TEM and immediately afterwards reassessed on the force platform.

DETAILED DESCRIPTION:
Aging is considered a dynamic and progressive process, in which morphological, functional and biochemical changes occur. One of the factors associated with old age is the decrease in the ability to balance posture and the high risk of falls. The literature brings the benefits of physical exercise in improving balance and preventing falls. However, few studies point to the benefits of flexibility techniques and their relationship with balance. The objective of this research is to evaluate the immediate effect of the muscle energy technique (TEM) on postural control responses in the elderly and young adults. The sample will be selected for convenience, with 50 participants of both sexes, young people between 18 and 35 years old and elderly people between 60 and 85 years old. Evaluation of postural control will be performed through the force platform during the unipodal and semi-tandem balance tests (2 repetitions of 30 seconds each, with rest of 30 seconds between them). The main parameters of postural control will be calculated using the pressure center derivative. After the balance tests, the participants will be submitted to TEM and immediately afterwards reassessed on the force platform. An analysis of variance will be used to compare the effects between groups (young versus elderly) and intervention (pre- and post-TEM) and the effects of interaction on the main variables of postural control. A beneficial effect of TEM is expected, especially in the elderly group. The results found in this study will contribute to the use of TEM and the increase of relevant clinical information to benefit the ability to balance in the elderly, in order to reduce the risk of falls.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in a study on a voluntary basis;
* Aged between 18 and 35 years old for young adults and over 60 years old up to 85 years old for elderly people;
* Being physically independent;
* Not practicing regular physical activity as recommended by the ACSM 3 to 5 times a week with moderate and severe;
* Cognitive status> 18 in the Mini-Mental State Examination.

Exclusion Criteria:

* Elderly with cognitive changes detectable by the Mini Mental State Examination (MMSE);
* A score lower than the score predicted for their level of education;
* Self-reported injuries;
* Falls in the last year;
* Musculoskeletal disorders;
* Systemic neurological-degenerative disease;
* Severe labyrinthitis and chronic diseases of the cardiovascular or respiratory system.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Balance | Baseline
  Balance measured by a Force platform

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Functional Assessment and Human Motor Performance (LAFUP), Londrina, Paraná, Brazil

REFERENCES:
- [Background] MINATTO et al. Idade, maturação sexual, variáveis antropométricas e composição corporal: influências na flexibilidade. Rev Bras Cineantropom Desempenho Hum. 2010;12(3):151-8.
- [Background] FRYER G, FOSSUMC. Therapeutic mechanisms underlying muscle energy approaches. In: Fernandez-de-las-Penas C, Arendt-Nielsen Lars, Gerwin R D editor(s). Tension-Type and Cervicogenic Headache: Pathophysiology, Diagnosis, and Management. Sudbury, MA: Jones and Bartlett Publishers,2010.
- [Background] Horak FB, Henry SM, Shumway-Cook A. Postural perturbations: new insights for treatment of balance disorders. Phys Ther. 1997 May;77(5):517-33. doi: 10.1093/ptj/77.5.517. PMID 9149762
- [Background] CHAITOW L. Técnicas de energia muscular. São Paulo: Manole; 2001
- [Background] Magnusson SP, Simonsen EB, Aagaard P, Dyhre-Poulsen P, McHugh MP, Kjaer M. Mechanical and physical responses to stretching with and without preisometric contraction in human skeletal muscle. Arch Phys Med Rehabil. 1996 Apr;77(4):373-8. doi: 10.1016/s0003-9993(96)90087-8. PMID 8607762
- [Background] Lariviere C, Gagnon D, Loisel P. The comparison of trunk muscles EMG activation between subjects with and without chronic low back pain during flexion-extension and lateral bending tasks. J Electromyogr Kinesiol. 2000 Apr;10(2):79-91. doi: 10.1016/s1050-6411(99)00027-9. PMID 10699556
- [Background] Shultz S, Averell K, Eickelman A, Sanker H, Donaldson MB. Diagnostic accuracy of self-report and subjective history in the diagnosis of low back pain with non-specific lower extremity symptoms: A systematic review. Man Ther. 2015 Feb;20(1):18-27. doi: 10.1016/j.math.2014.08.002. Epub 2014 Aug 29. PMID 25231775
- [Background] Bertolucci PH, Brucki SM, Campacci SR, Juliano Y. [The Mini-Mental State Examination in a general population: impact of educational status]. Arq Neuropsiquiatr. 1994 Mar;52(1):1-7. Portuguese. PMID 8002795
- [Background] Baecke JA, Burema J, Frijters JE. A short questionnaire for the measurement of habitual physical activity in epidemiological studies. Am J Clin Nutr. 1982 Nov;36(5):936-42. doi: 10.1093/ajcn/36.5.936. PMID 7137077
- [Background] Voorrips LE, Ravelli AC, Dongelmans PC, Deurenberg P, Van Staveren WA. A physical activity questionnaire for the elderly. Med Sci Sports Exerc. 1991 Aug;23(8):974-9. PMID 1956274
- [Background] Province MA, Hadley EC, Hornbrook MC, Lipsitz LA, Miller JP, Mulrow CD, Ory MG, Sattin RW, Tinetti ME, Wolf SL. The effects of exercise on falls in elderly patients. A preplanned meta-analysis of the FICSIT Trials. Frailty and Injuries: Cooperative Studies of Intervention Techniques. JAMA. 1995 May 3;273(17):1341-7. PMID 7715058
- [Background] Adaptação do Habitual Physical Activity Questionnaire (Baecke), versão modificada, para a população portuguesa. Maria Celeste Bastos Almeida; José Luís Pais Ribeiro.
- [Background] Camargos FF, Dias RC, Dias JM, Freire MT. Cross-cultural adaptation and evaluation of the psychometric properties of the Falls Efficacy Scale-International Among Elderly Brazilians (FES-I-BRAZIL). Rev Bras Fisioter. 2010 May-Jun;14(3):237-43. English, Portuguese. PMID 20730369
- [Background] Wells KF, Dillon EK. The sit and reach: a test of back and leg flexibility. Research Quarterly for Exercise and Sport, Washington, 1952, 23:115-118.
- [Background] Fitness Canada. Canadian Standardized Test of Fitness (CSTF) Operations Manual. 3rd Ed. Ottawa: Fitness and Amateur Sport, Canada, 1986
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946